CLINICAL TRIAL: NCT04473716
Title: Neoadjuvant Toripalimab and Paclitaxel/Cisplatin on Pathological Response in Oral Squamous Cell Carcinoma Patients: A Single-arm Phase I Trial
Brief Title: Neoadjuvant Toripalimab and Paclitaxel/Cisplatin on Pathological Response in Oral Squamous Cell Carcinoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Illuminate trial
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Oral Cancer; Induction Chemotherapy; Programmed Cell Death 1 Inhibitor; Inductive Therapy
MeSH Terms: conditions — Mouth Neoplasms | interventions — toripalimab; Injections; Paclitaxel; Cisplatin; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy with Toripalimab, Paclitaxcel and Cisplatin (Experimental): Pre-operative neoadjuvant therapy will be used with the combination of immune checkpoint inhibitor of Toripalimab, and chemotherapy agents of paclitaxcel and cisplatin in patients with locally advanced OSCC. After inductive therapy, the patients will receive radical surgery and post-operative radiotherapy/chemoradiotherapy.
  Interventions: Drug: Toripalimab; Drug: Paclitaxcel; Drug: Cisplatin; Procedure: Radical surgery; Radiation: Post-operative radiotherapy/chemoradiotherapy

INTERVENTIONS:
Drug: Toripalimab — Neoadjuvant therapy with Toripalimab of 240mg, iv, qd, on day 1, 22
  Other Names: Toripalimab for Injection
Drug: Paclitaxcel — Neoadjuvant therapy with Paclitaxcel of 260mg/m2, iv, qd, on day 1, 22
  Other Names: Paclitaxel for Injection (Albumin Bound)
Drug: Cisplatin — Neoadjuvant therapy with Cisplatin of 75mg/m2, iv, qd, on day 1, 22
  Other Names: Cisplatin for Injection
Procedure: Radical surgery — Radical surgery will be performed on the 43th-48th after initiation of inductive therapy.
Radiation: Post-operative radiotherapy/chemoradiotherapy — Post-operative radiotherapy/chemoradiotherapy will be performed within 1.5 months after radical surgery, depending on the post-operative pathological diagnosis.

SUMMARY:
The aim of this study is to use the combination of immune checkpoint inhibitor of Toripalimab, and chemotherapy agents of TP, as a neoadjuvant therapy to treat the patients with locally advanced OSCC, followed with radical surgery and post-operative radiotherapy/chemoradiotherapy, the major pathological response and safety will be evaluated as the primary surrogate endpoints, the 2-year survival rate and local recurrence rate will be the second endpoints.

DETAILED DESCRIPTION:
In patients with locally advanced oral squamous cell carcinoma (OSCC), comprehensive treatment is recommended, including surgery, radiotherapy, chemotherapy and others. Pre-operative neoadjuvant therapy can reduce tumor burden, increase organ preservation rate, and reduce distant metastasis rate. Pre-operative neoadjuvant therapy with paclitaxcel and cisplatin (TP) has been used as one of recommended protocols in patients with locally advanced head and neck squamous cell caricnoma, including OSCC. Anti-PD1/PD-L1 immunotherapies have achieved exciting clinical outcomes in several malignancies, such as lung cancer, breast cancer, and so on. Recently, pre-operative neoadjuvant therapy with combination of immunotherapy and chemotherapy agents has been used with good pathological response, which might transfer to good clinical prognosis in patients with malignancies. However, pre-operative neoadjuvant therapy with combination of anti-PD1 and TP in OSCC patients has not been reported. The innovation of this study is the combination of immune checkpoint inhibitor of Toripalimab, and chemotherapy agents of TP, as a neoadjuvant therapy to treat the patients with locally advanced OSCC, followed with radical surgery and post-operative radiotherapy/chemoradiotherapy, the major pathological response and safety will be evaluated as the primary surrogate endpoints, the 2-year survival rate and local recurrence rate will be the second endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Eastern cooperative oncology group performance status (ECOG PS) score: 0-1 points
* Pathological diagnosis of oral squamous cell carcinoma (including tongue, gums, cheeks, mouth floor, hard palate, posterior molar region)
* Clinical stage of III/IVA (AJCC 2018)
* Blood routine: white blood cells > 3,000/mm3, hemoglobin > 8g/L, platelets > 80,000/mm3
* Liver function: Alanine Transaminase/Aspartate Transaminase <2.5 times the upper limit of normal, bilirubin <1.5 times the upper limit of normal
* Renal function: serum creatinine <1.5 times the upper limit of normal
* Sign the informed consent

Exclusion Criteria:

* There are still unresolved toxic reactions above CTCAE level 2 caused by previous anti-cancer treatment
* Grade 3-4 allergic reactions to Toripalimab, paclitaxcel or cisplatin
* Active severe clinical infection (> CTCAE 5.0 version 2 infection)
* Difficult to control hypertension or cardiovascular disease with clinical significance (such as activity)-such as cerebrovascular accident (< 6 months before treatment), myocardial infarction (< 6 months before treatment), unstable angina, New York Cardiology Society (NYHA Appendix 5) congestive heart failure grade II or above, or severe arrhythmia that cannot be controlled with drugs or has potential impact on experimental treatment
* Chronic diseases requiring immunotherapy or hormone therapy
* Women during pregnancy or lactation
* Participated in other clinical studies within 30 days before enrollment
* Other circumstances that the investigator thinks are not suitable for participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Major pathological response | One year
  Major pathological response is based on the pathological examination on the post-operative specimens after neoadjuvant therapy.

SECONDARY OUTCOMES:
2-year overall survival | Two years
  The overall survival time refers to the time from initiating inductive therapy to death due to any cause.
2-year tumor recurrence rate | Two years
  The tumor recurrence rate is calculated using the number of patients with tumor recurrence divided by the total number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lai-ping Zhong, MD, PhD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Ninth People's Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Huang Y, Sun J, Li J, Zhu D, Dong M, Dou S, Tang Y, Shi W, Sun Q, Zhao T, Zhou Z, Zhou X, Liu Y, Li J, Zhu G, Zhang D, Chen Y, Zhu Q, Ju W, Zhong L. Neoadjuvant immunochemotherapy for locally advanced resectable oral squamous cell carcinoma: a prospective single-arm trial (Illuminate Trial). Int J Surg. 2023 Aug 1;109(8):2220-2227. doi: 10.1097/JS9.0000000000000489. PMID 37288582